CLINICAL TRIAL: NCT04279431
Title: Follow-up of MTBI Patients Discharged from the ED Using Standard Clinical Triage Including BrainScope One
Acronym: MEDO
Status: Active, not recruiting | Type: Observational
Sponsor: BrainScope Company, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MEDO-40
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: TBI (Traumatic Brain Injury); Concussion, Brain; MTBI - Mild Traumatic Brain Injury; Closed Head Injury
Keywords: BrainScope; Closed Head Injury; Concussion; EEG Evaluation; Cognitive Evaluation; Concussion Symptom Inventory; mTBI
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Head Injuries, Closed | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- SIC Negative: Subjects will include males and females ranging from ages 18 to 85 who are admitted to the ED with a traumatic, closed head injury within 3 days of injury. Subject will undergo site standard clinical ED evaluation and a BrainScope evaluation. The SIC negative group are those patients who obtain a 'Negative' result on the BrainScope One Structural Injury Classifier (SIC) algorithm.
  Interventions: Device: EEG Recording; Other: Neurocognitive Tests; Other: Clinician Evaluation; Other: 22-item CSI
- SIC Positive/Equivocal: Subjects will include males and females ranging from ages 18 to 85 who are admitted to the ED with a traumatic, closed head injury within 3 days of injury. Subject will undergo site standard clinical ED evaluation and a BrainScope evaluation. The SIC positive group are those patients who obtain a 'Positive' or 'Equivocal' result on the BrainScope One SIC algorithm.
  Interventions: Device: EEG Recording; Other: Neurocognitive Tests; Other: Clinician Evaluation; Other: 22-item CSI

INTERVENTIONS:
Device: EEG Recording — EEG recording acquired on BrainScope One device.
Other: Neurocognitive Tests — Cognitive performance tests performed on BrainScope One device.
Other: Clinician Evaluation — Clinician evaluation performed as part of standard of care at the clinical site.
Other: 22-item CSI — Self assessed 22-item Concussion Symptom Inventory (CSI).

SUMMARY:
The purpose of the study is to validate the clinical outcome in patients with closed head injuries (GCS 14-15, ages 18-85) who are being evaluated for head trauma, integrating the BrainScope One structural injury classifier (SIC) algorithm, with focus on SIC negative classification. In addition, to assess functional impairment (concussion) in these patients, results from Brain Function Index (BFI) or Concussion Index (CI) algorithms will be used for analysis.

DETAILED DESCRIPTION:
BrainScope One incorporates brain electrical activity (EEG, a proven electrophysiological core technology) and other multimodal assessment capabilities in a portable, point-of-care, non-invasive device containing algorithms designed to improve early identification, staging, and optimization of treatment for head injured patients (GCS 13-15) who are suspected of a brain injury. Structural Injury Classifier (SIC) provides objective results that indicate the likelihood of a structural brain injury being present, potentially visible on CT Scan. Brain Function Index (BFI) provides an objective measurement to determine the likelihood and severity of brain function impairment such as that seen in concussion/mTBI. The BFI is presented as a percentile compared to a normal corresponding population. Lastly, the Concussion Index (CI) was derived in the most recent BrainScope concussion assessment clinical study, and it is defined as a multivariate, multimodal index to assess the presence and severity of concussion and has been demonstrated to reliably reflect change over time.

The present study population targets those patients who sustained a head injury, have high GCS scores (14-15) and present mild symptoms, for whom the suspicion of structural brain injury is therefore low. Having a rapid, reliable, and sensitive assessment tool to aid in the triage of patients who are suspected of a traumatically induced structural brain injury could aid in appropriate and timely diagnosis and subsequent medical care. It may also result in more appropriate utilization of medical imaging (potentially having associated health risks) and reductions in hospitalizations. Patients discharged from the ED who were deemed to not require a CT scan will be followed-up for outcome.

ELIGIBILITY:
* Inclusion Criteria:

  1. Patient can be of any gender;
  2. Patient must be admitted to the ED with a traumatic closed head injury within 72 hours of injury;
  3. Patient's Age must be ≥18 and <86 years old at time of enrollment;
  4. Patient must be Glasgow Coma Scale (GCS) 14-15 at time of BrainScope evaluation (even if GCS was lower prior to arrival e.g. at time of injury).
* Exclusion Criteria:

  1. Patients with forehead, scalp, earlobe or skull abnormalities or other conditions that would prevent correct application of the electrode headset;
  2. Patients with Dementia, Parkinson's Disease, Multiple Sclerosis, brain tumors, history of brain surgery, evidence of acute psychosis or history of stroke with neurological deficit within the last year;
  3. Patients on anti-platelets, anti-coagulants, other than aspirin, currently receiving dialysis or in end-stage renal disease or current condition is "critical" in the opinion of the investigator;
  4. Patients with active fever defined as greater than 100oF or 37.7oC;
  5. Patients suffering from an open head injury or have suffered multi-trauma which requires hospitalization (for injuries not related to the head injury)
  6. Patients requiring advanced airway management (i.e. mechanical ventilation);
  7. Patients currently receiving procedural sedation medications (e.g. benzodiazepine, anesthetic, NMDA receptor antagonist, or opioid agonist) Note: patient can be enrolled when they are no longer obtunded and have the capacity to consent;
  8. Pregnant women and prisoners;
  9. Patients who have had a Head CT scan for current traumatic injury event prior to screening.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An estimated total of 660 patients (with target of 330 SIC negative patients) who are suspected of a traumatic, closed head injury within 3 days of injury, will be recruited from patients who enter the participating Hospital ED's as clinical sites for this study. Potential study subjects will be identified by the research staff based on the stated inclusion and exclusion criteria to determine their eligibility. Once identified, the research staff will recruit the subject for the study through an informed consent process. Participation in the study will not interfere with standard of care at the clinical sites.
Sampling Method: Non-Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2020-05-25 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical utility of integration of BSC SIC into the triage of closed head injured patients. | 30 days
  Demonstrate the accuracy of the BrainScope Structural Injury Classifier (SIC) negative findings through repeated follow ups of those patients discharged from the ED without receiving a CT scan, as determined by the ED physician.

SECONDARY OUTCOMES:
High NPV adds confidence to the clinical decision not to scan when the BrainScope SIC is negative | After enrollment closure
  For those who were BSC SIC negative and who are referred to CT due to clinician's decision, CT results will be obtained to assess the accuracy of BrainScope finding, this will allow an estimate of NPV.
Higher specificity in BSC SIC compared to Nexus II and CCHR could result in decrease of referral for unnecessary CT scans due to higher specificity. | After enrollment closure
  Compare accuracy of Nexus II and CCHR Imaging rules to BrainScope in predicting true negatives
To correlate BFI and CI to the severity and duration of concussive symptom burden (measured by CSI) | After enrollment closure
  The BFI/CI can help to inform the clinical decision on the likely of concussion at the time of injury in the ED environment and predict prolonged recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie S Prichep, Ph.D., Study Director — BrainScope Company, Inc.
Locations (7):
- United States (7):
  - Wayne State University - Detroit Receiving Hospital, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Wayne State University - Sinai Grace Hospital, Detroit, Michigan
  - Beaumont Hospital, Royal Oak, Michigan
  - Beaumont Hospital, Troy, Michigan
  - Washington University - Barnes Jewish Hospital, St Louis, Missouri
  - El Paso Medical Center, El Paso, Texas

IPD SHARING:
Plan to Share IPD: No